CLINICAL TRIAL: NCT02055807
Title: Role of Lung Ultrasound Imaging in the Comparison of Two Mechanical Ventilation Strategies During Laparotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.293
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Atelectasis
Keywords: Atelectasis; Ultrasound; Recruitment maneuver; Positive end-expiratory pressure
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEP and recruitment maneuvers (Experimental): A PEEP of 7 cm H2O will be applied starting after intubation until the end of surgery. Recruitment maneuvers (continuous positive pressure of 30 cm H20 for 30 seconds) will be initiated following intubation and repeated every 30 minutes during surgery and immediately prior to extubation. Lung ultrasound examinations will be performed at different time-points immediately before surgery, during surgery under general anesthesia and after surgery in the recovery room to detect and monitor atelectasis.
  Interventions: Other: PEEP and recruitment maneuvers
- ZEEP (Zero end-expiratory pressure) (Active Comparator): No PEEP nor recruitment maneuvers will be used during surgery. Lung ultrasound examinations will be performed at different time-points immediately before surgery, during surgery under general anesthesia and after surgery in the recovery room to detect and monitor atelectasis.
  Interventions: Other: ZEEP (no PEEP nor recruitment maneuver)

INTERVENTIONS:
Other: PEEP and recruitment maneuvers
  Arms: PEEP and recruitment maneuvers
Other: ZEEP (no PEEP nor recruitment maneuver)
  Arms: ZEEP (Zero end-expiratory pressure)

SUMMARY:
The use of positive end-expiratory pressure (PEEP) and recruitment maneuvers during laparotomy will limit the development of atelectasis and therefore improve the aeration score.

DETAILED DESCRIPTION:
Postoperative pulmonary complications contribute to the morbidity of surgical patients. During general anesthesia, up to 90% of patients will develop atelectasis, which is thought to be a major contributing factor to their development. The adjustment of ventilator settings to prevent the occurrence of atelectasis and reduce pulmonary complications remains controversial. Despite the use of similar mechanical ventilation strategies, two recent studies (IMPROVE, PROVHILO) involving 1300 patients diverged in their conclusions regarding the impact of these strategies in the prevention of pulmonary complications. In these studies, the absence of imagery to assess the pulmonary end-result of the different ventilation strategies complicates the interpretation of their results.

On arrival in the operating theatre, each patient will undergo a baseline lung ultrasound examination. The anesthetic technique and monitoring will be standardized. The radial artery will be cannulated after induction of anesthesia for blood gas monitoring. Ventilator settings will be adjusted according to randomization.

A second lung ultrasound examination will be performed 5 minutes following induction of general anesthesia. In the PEEP group, a lung ultrasound examination will be performed immediately following the first recruitment maneuver. A lung ultrasound examination will also be performed at the end of surgery before emergence of general anesthesia.

Fifteen minutes after arrival in the recovery room, a last lung ultrasound examination will be performed. Fraction of inspired oxygen (FiO2) and vital signs will be recorded during each ultrasound examination. Arterial blood samples will be collected simultaneously. The aeration score will be calculated for each lung ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Scheduled for surgery by laparotomy (expected to last at least 2 hours)
* American Society of Anesthesiologists classification: physical status 1-3

Exclusion Criteria:

* Previous thoracic procedure (thoracic drain, thoracotomy, thoracoscopy)
* Contraindication to the placement of an arterial line
* Very severe chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Lung aeration | Post-induction to pre-emergence of anesthesia - Day 0
  Compare lung aeration between two different mechanical ventilation strategies (with or without PEEP and recruitment maneuvers) using ultrasound imaging and a four point aeration score (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation).

SECONDARY OUTCOMES:
Re-aeration following recruitment maneuvers | Prior and after the first recruitment maneuver during general anesthesia - Day 0
  Assess lung re-aeration following a recruitment maneuver by ultrasound imaging (lung aeration score pre/post the first recruitment maneuver during general anesthesia).
Atelectasis secondary to induction | Lung aeration score prior and after intubation - Day 0
  Estimate development of atelectasis secondary to intubation.
Atelectasis secondary to extubation | Lung aeration score prior and after extubation - Day 0
  Estimate development of atelectasis secondary to extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Genereux V, Chasse M, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Effects of positive end-expiratory pressure/recruitment manoeuvres compared with zero end-expiratory pressure on atelectasis during open gynaecological surgery as assessed by ultrasonography: a randomised controlled trial. Br J Anaesth. 2020 Jan;124(1):101-109. doi: 10.1016/j.bja.2019.09.040. Epub 2019 Nov 14. PMID 31733807